CLINICAL TRIAL: NCT04418856
Title: Light Therapy to Treat Cancer-related Fatigue, Sleep Problems, Depression and Cognitive Impairment Among Breast Cancer Patients.
Brief Title: The Effects of Light Therapy to Treat Cancer-related Side Effects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reykjavik University (Other)
Collaborators: The Icelandic Research Fund (Unknown)
Responsible Party: Principal Investigator, Dr. Heiddis B Valdimarsdottir, Professor, Reykjavik University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VSN-18-199
Record Dates: First submitted 2020-05-05; First posted 2020-06-05 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer; Circadian Rhythms; Fatigue; Sleep Disturbance; Cognitive Impairment; Inflammatory Response; Depression
Keywords: Breast cancer; Light therapy; Cancer related side effects; Circadian rhythms; Inflammatory markers
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Parasomnias; Cognitive Dysfunction; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Experimental light: Breast cancer surgery and chemotherapy (Experimental): Exposed to experimental systematic light exposure for 30 minutes each morning from the time of breast cancer surgery until the end of the chemotherapy treatment
  Interventions: Device: Light Glasses (Experimental)
- Comparison Light:Breast cancer surgery and chemotherapy (Active Comparator): Exposed to comparison systematic light exposure for 30 minutes each morning from the time of breast cancer surgery until the end of the chemotherapy treatment
  Interventions: Device: Light Glasses (Comparison)
- Experimental light: Breast cancer surgery and no chemotherapy (Experimental): Exposed to experimental systematic light exposure for 30 minutes each morning for four weeks starting at the time of breast cancer surgery
  Interventions: Device: Light Glasses (Experimental)
- Comparison light: Breast cancer surgery and no chemotherapy (Active Comparator): Exposed to experimental systematic light exposure for 30 minutes each morning for four weeks starting at the time of breast cancer surgery
  Interventions: Device: Light Glasses (Comparison)
- Healthy control group (No Intervention): The healthy control group and the breast cancer patients undergo the same assessments (questionnaires, neuropsychological assessments and actigraphy) at the same time points

INTERVENTIONS:
Device: Light Glasses (Experimental) — The light glasses emit light from LEDs at a distance of 15 millimeters (15mm, 0.015.) from the eye. The device is classified as safe for the eyes in accordance with the international standard IEC 62471 and complies with the United States of America's FCC marking, and is designed to be worn on the participant's head, similar to a pair of glasses. For safety purposes, the light glasses do not contain UV or infra-red light.
  Arms: Experimental light: Breast cancer surgery and chemotherapy; Experimental light: Breast cancer surgery and no chemotherapy
Device: Light Glasses (Comparison) — The light glasses emit light from LEDs at a distance of 15 millimeters (15mm, 0.015.) from the eye. The device is classified as safe for the eyes in accordance with the international standard IEC 62471 and complies with the United States of America's FCC marking, and is designed to be worn on the participant's head, similar to a pair of glasses. For safety purposes, the light glasses do not contain UV or infra-red light.
  Arms: Comparison Light:Breast cancer surgery and chemotherapy; Comparison light: Breast cancer surgery and no chemotherapy

SUMMARY:
Severe fatigue, depression, sleep problems and cognitive impairment are the most commonly reported side effects of cancer treatment. These aversive side effects are hypothesized to be related to the disruption of circadian rhythms associated with cancer and its treatment. Exposure to Bright White Light (BWL) has been found to synchronize the circadian activity rhythms but research with cancer patients has been scarce. Therefore, the proposed randomized control trial (RCT) will test if systematic light exposure (sLE) will minimize overall levels of cancer-related fatigue (CRF), depression, sleep problems and cognitive impairment among breast cancer patients undergoing breast cancer treatment (i.e., surgery, chemotherapy). SLE incorporates the delivery of harmless UV-protected BWL or Dim White Light (DWL - standard comparison in light studies) delivered to patients by using special glasses for 30 minutes each morning, during their treatment. The proposed study, including a delineated comparison condition, will investigate the effects of BWL on CRF, sleep, depression, cognition, circadian rhythms, and inflammation markers among patients undergoing breast cancer treatment. The proposed RCT could have major public health relevance as it will determine if an easy-to-deliver, inexpensive, and low patient burden intervention reduces common side effects (e.g., CRF, depression, cognitive impairment) of cancer treatment (i.e., surgery, chemotherapy).

Aim 1 - Assess whether Bright White Light (BWL) compared with Dim White Light (DWL) among breast cancer patients undergoing breast cancer treatment will minimize overall levels of CRF, depression, sleep problems, and cognitive impairment during and after breast cancer treatment, compared to healthy controls.

Aim 2 - Determine whether the BWL intervention affects cortisol rhythms, circadian activity rhythms, melatonin rhythms, and inflammation markers that have been identified as correlates/causes of cancer-related side effects (e.g., CRF, depression, sleep problems).

Aim 3 - Exploratory: Explore whether the effects of BWL compared to DWL on the cancer-related side effects (e.g., CRF, cognitive impairment) are mediated by the beneficial effects of the BWL in synchronizing circadian rhythms.

Aim 4 - Exploratory: Explore potential moderators of the intervention including seasonality, chronobiology, personality, and social factors.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer Patients: Newly diagnosed patients with stages 1 to 3 breast cancer scheduled to undergo surgery (without chemotherapy) and newly diagnosed patients with stages 1 to 3 breast cancer scheduled to undergo both surgery and chemotherapy.
2. Healthy controls: never received a cancer diagnosis

Exclusion Criteria:

* Stage 3B breast cancer, inflammatory or stage 4 breast cancer; under age 18; pregnancy; pre-existing anemia (Hb <10gm/dl); history of bipolar disorder or mania (which are contra-indications for BWL treatment); and any other physical or psychological impairments (e.g., sleep disorder diagnosis) which could limit participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 240 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
FACIT-Fatigue Scale | Up to 14 months
  The FACIT-Fatigue Scale is an outcome measure of fatigue consisting of 13 items on a four point Likert scale about fatigue levels during usual daily activities over the past 7 days. The scale has excellent test-retest reliability (r = 0.90) and internal consistency reliability (α= 0.93-0.95).
Pittsburgh Sleep Quality Index | Up to 14 months
  The Pittsburgh Sleep Quality Index assesses sleep quality. The scale consists of 19 self-rated items, divided into seven components. The scores ranges from 0-21, with lower scores indicating better sleep quality. The scale has the test-retest reliability of r=.85 and estimated internal consistency of α=.80.
The Center for Epidemiological Studies Depression Scale | Up to 14 months
  The Center for Epidemiological Studies Depression Scale (CES-D) measures depression symptoms. The 20 items scores range from 0 - 60, with higher scores indicating greater depressive symptoms. Internal consistency for women undergoing breast cancer treatment is estimated to be α=.89 and α=.90 for healthy comparison group.
PROMIS cognitive function and cognitive abilities | Up to 14 months
  PROMIS® (Patient-Reported Outcomes Measurement Information System) cognitive function and cognitive abilities 8a consist of 8 self-report item rated on a five point Likert scale ranging from "never" to "very often" on the Cognitive Function scale and "not at all" to "very much" on the Cognitive Abilities scale. Both PROMIS item banks show good psychometric properties, such as a high internal consistency (α =.94 for each).
The Rey 15-Item Memory Test | Up to 14 months
  The Rey 15-Item Memory Test evaluates short-term memory along with long-term memory. The test consists of series of 15 common words and the subject freely expressing the words retained. Afterward, another list of 15 unrelated words are given and the task of the subject is to repeat the original list of 15 words and then to repeat it after 30 minutes. RAVLT has good internal consistency (α=.80) and adequate convergent and divergent validity.
The Digit Span test | Up to 14 months
  The Digit Span test assesses working memory and immediate auditory recall. It is a part of the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV). The test has two subsections: Digits forwards and Digits backwards, each containing eight items. The task of the participants is to repeat the sequence of numbers the examiner reads for them, either repeat exactly what the examiner said or reverse it. Its reliability and validity is considered to be good, with internal consistency of 0.79, test-retest reliability of 0.77 and split-half reliability of 0.88.
The Stroop task | Up to 14 months
  The Stroop task assesses selective attention, or the ability of the participant to block out irrelevant stimuli. The first subtask consists of reading color names (yellow, red, green and blue) written in black ink as fast as possible, in order to measure the reading and psychomotor speed of the participants. The second subtask consists of naming colored pads and in the third subtask the participants say the font color in which the color names are written in, which do not necessarily match. Stroop has been found to be stable across the one- and two week period with a test-retest coefficient of 0.83 for the Word task, 0.74 for the Color task and 0.67 for the Color Word task.
The Trail Making test | Up to 14 months
  The Trail Making Test (TMT) consists of two parts: TMT A and B. TMT A measures visual search and psychomotor speed, whereas TMT B measures divided attention, cognitive flexibility and working memory. In TMT A, the task of the participants is to draw a line as quickly as they can between 25 circles in the correct order without lifting their pencil, with each circle containing a number from 1-25 presented in an random array. In TMT B, the task of the participants is to draw a line between randomly arranged encircled numbers from 1 to 13 and letters from A to L, in the correct sequence while alternating between letters and numbers, as quickly and accurately as they can. Test-retest reliability of 0.79 has been found for part A and 0.89 for part B.
Psychomotor Vigilance task | Up to 14 months
  Psychomotor vigilance task (PVT) measures alertness and vigilant attention and is considered to be the gold standard measure of neurobehavioral effects of circadian misalignment and sleep loss. In PVT participants are instructed to attend to a red rectangular box on a computer screen and to respond to a yellow stimulus counter inside the box. PVT gives information about accuracy and reaction time. The test has shown good psychometric properties, such as high reliability, with intra-class correlations assessing test-retest reliability above 0.8.
The automated Operation Span task | Up to 14 months
  The automated operation span task (aOSPAN) measures working memory span and consists of solving math operations while remembering a set of letters in the correct order, in set sizes ranging from 2 to 5. The task starts with three practice trials. The aOSPAN gives information about accuracy and reaction time. AOSPAN has shown to be reliable across sessions (.83) and to load highly on the working memory capacity factor (.68).
The Word Fluency Test | Up to 14 months
  The Word Fluency test measures executive functioning and semantic abilities of the participants. This test is the Icelandic equivalent of the standard F-A-S test, employing the letters H and S since they are the most frequent letters in Icelandic. The initial part of the test consists of phonemic fluency tasks where the participants say as many words beginning with the letter H as fast as they possibly can in one minute, followed by the letter S. The latter part of the test measures semantic fluency where the participants are instructed to do the same but with animal names. The test has shown good internal consistency (α=.83) and test-retest reliability of .74.

SECONDARY OUTCOMES:
Salivary Cortisol | Up to 14 months
  Salivary Cortisol: A commercial chemiluminescence immunoassay (CLIA) will be used to analyze the saliva samples, with a lower detection limit of 0.41 nmol/L. Inter- and intra-assay coefficients of variance are <10% across the expected range of cortisol levels. The following parameters will be calculated and used in analyses: 1) the cortisol awakening response (the rise in cortisol from waking to 30 minutes post-waking), 2) nocturnal cortisol, and 3) the diurnal cortisol slope.
Urinary Melatonin | Up to 14 months
  Production of pineal melatonin can be inferred from urinary 6 sulfatoxymelatonin (major metabolite of melatonin in urine). Urinary aMT6s (ng/mg Creatinine) will be measured by a competitive ELISA kit. Total excretion of aMT6s is calculated by multiplying the assayed concentration by the volume of urine voided. The aMT6s profiles will be analyzed using cosinor analysis, which is based on the least square approximation of the time series using a cosine function with a period of 24 h. The following parameters will be calculated: 1) acrophase time: time of the peak aMT6s concentration; 2) mesor: mean aMT6s value for all the samples included in the cosinor analysis and 3) amplitude: difference between the mesor and the peak aMT6s level.
Circadian Activity Rhythms | Up to 14 months
  Circadian Activity Rhythms (CAR) will be recorded with a wrist actigraphy or ActTrust. ActTrust generates the the following three CAR parameters: 1) Amplitude (peak or maximum of the curve, with a lower amplitude indicating a less rhythmic rhythm); 2) Acrophase (time of day of the peak activity, with a later time indicating more phase-delay); and 3) Mesor (half-way between minimum and maximum of the curve, a circadian rhythm-adjusted mean of the daily activity).
Connor-Davidson Resilience Scale | Up to 14 months
  Connor-Davidson Resilience Scale (CD-RISC-10) is a 10 item ordinal scale rated on a 5-point (0-4) scale with higher scores reflecting greater resilience. It is meant to measure one's ability to "bounce-back" and propensity for adaptability. The scale has excellent Internal Consistency, α=.85.
Positive and Negative Affect Schedule | Up to 14 months
  Positive and Negative Affect Schedule (I-PANAS-SF) shorter version is a self-report affect scale that measures positive and negative feelings on a 5-point Likert scale, consisting of five positive stated and five negative stated questions, in total 10 questions. The scale has good internal reliability, or α=.82.
The Credibility/Expectation Questionnaire | Up to 14 months
  The Credibility/Expectation Questionnaire (CEQ) consists of 5 items listed on a 10-point self-report scale that measures treatment credibility and expectancy in clinical outcome studies. The scale has high internal consistency within the two factors, credibility α=.81 and expectation α=.90, and good test-retest reliability.
Godin-Shephard Leisure-Time Physical Activity Questionnaire | Up to 14 months
  Godin-Shephard Leisure-Time Physical Activity Questionnaire (GSLTPAQ)/Godin-Shephard Leisure-Time Exercise Questionnaire (GLTEQ) consists of three self-report questions were respondents rates their weekly leisure activity, such as how often and how strenuous they typically exercise. The leisure score index is obtained by the multiplying the frequency of each score with a corresponding Metabolic Equivalent of Task (MET) value, dividing the total score in three categories: active (24 units or more), moderately active (14 to 23 units) and less substantial or low benefits (14 units or less).
The reduced Horne & Östberg Morningness-Eveningness Questionnaire | Up to 14 months
  The reduced Horne & Östberg Morningness-Eveningness Questionnaire (rMEQ) is a self-report questionnaire consisting of 5 questions that assess chronotypes, where a higher score suggests a morningness chronotype. Its internal consistency has been estimated to be α=.69 - .78.
Severity of cancer symptoms | Up to 14 months
  MD Anderson Symptom Inventory (MDASI) is a symptom-specific patient-reported outcome instrument that consists of 19 questions developed to direct access symptoms experienced by cancer patients and how much they interfere with daily living. The inventory has a good internal consistency and test-retest reliability of α= ≥ .84 and intraclass correlation for all subscales ≥ .76.
SF-12 | Up to 14 months
  SF-12 consists of 12 items that measure health related quality of life, both physical and mental wellbeing, and is the shorter form of the SF-36 questionnaire. A study among breast cancer survivors found an internal consistency of α > .85.
The Life Events Checklist | Up to 14 months
  The Life Events Checklist (LEC) assesses exposure to 16 potentially traumatic events known to predict posttraumatic stress disorder or other posttraumatic difficulties. For each item, participants are asked whether the trauma exposure was direct or indirect. Its psychometric properties have proven decent, with good temporal stability and convergence with other established trauma history measures.
FACIT-TS-G | Up to 14 months
  FACIT-TS-G assesses how satisfied participants are with the treatment they received. In the current study we use 10 questions adapted to the Bright Light therapy, e.g. about potential side effects.
Hot Flashes | Up to 14 months
  In the current study we employ the Daily Patient questionnaire about Hot Flashes for female patients. The questionnaire consists of examples of how cancer patients in previous studies have defined symptoms of their hot flashes as mild, moderate, severe and very severe. The participants fill out a diary for a week, consisting of the number of hot flashes along with their severity for each day.
The Impact of Event Scale | Up to 14 months
  The Impact of Event Scale measures trauma related stress, that is cancer specific distress. It is a 22-item scale, divided up into three subscales; intrusion, avoidance and hyperarousal. Total scores range from 0-88, with higher scores suggesting more distress. High levels of internal consistency have been previously reported (Intrusion: α=.87 - 0.92, Avoidance: α=.84 - .85, Hyperarousal: α= .79 - .90). Test-retest correlation coefficients were reported moderate to high (Intrusion: .57 - .94, Avoidance: .51 - .89, Hyperarousal: .59 - .92).
The NCCN Distress Thermometer | Up to 14 months
  The NCCN Distress Thermometer and checklist is a widely used screening measure for distress in cancer patients. It consists of a distress thermometer where participants assess their distress on a scale from 0 to 10, were 0 indicates no distress and 10 extreme distress. Additionally, participants answer a problem checklist with several domains to identify what area of life distresses the participant.
The Social Constraints Scale | Up to 14 months
  The Social Constraints Scale (SCS) shorter version consists of 6 items, scored from "never" to "always" on a 4-point Likert scale. Social constraints assesses the perceived lack of social support from someone close to them, discouraging the cancer patient to express their cancer-related-emotions. The internal consistency of the scale has been shown to be adequate (α=.71 - .81).
Short Form of the Post-Traumatic Growth Inventory | Up to 14 months
  Short Form of the Post-Traumatic Growth Inventory (PTGI-SF) is a 10-item ordinal scale used to assess positive outcomes after a traumatic event. The scale has excellent internal consistency (α=.86) and appears to have utility in determining how successful individuals are in reconstructing or strengthening their perceptions of self, others, and the meaning of events.
The Generalized Anxiety Disorder | Up to 14 months
  The Generalized Anxiety Disorder-7 (GAD-7) is a 7-item measure used to screen for general anxiety disorder and its severity. The scale is on 4-point Likert scale ("not at all" to "several days") and the score ranges from 0-21, with higher scores indicating more severe anxiety. Its internal consistency is estimated excellent (α=.92).
The Perceived Stress Scale | Up to 14 months
  The Perceived Stress Scale (PSS-10) is a 10-item scale used to measure stress. Each item on the list is rated on a 5-point Likert scale ranging from "never" to "very often". PSS-10 total score ranges from 0 to to 40, where a higher score indicates higher perceived stress. The scale has adequate reliability and validity.
Functional Assessment of Cancer Therapy-Breast | Up to 14 months
  Functional Assessment of Cancer Therapy-Breast version 4 (FACT-B v4) measures the multidimensional quality of life in breast cancer patients. The instrument consists of five subscales with 37 breast cancer-specific items. The scale demonstrates a good reliability, validity and internal consistency (α ≥ .70).
Sleep/wake activity | Up to 14 months
  Sleep/wake activity will be recorded with a wrist actigraphy or ActTrust. ActTrust actigraph generates the following seep/wake information: Percent sleep, number of awakenings per night, length of awakenings at night, percent wake, and napping behavior (number of naps defined as 10 minutes of inactivity; naptime).
Circadian Activity Rhythms - Amplitude | Up to 14 months
  Circadian Activity Rhythms (CAR) will be recorded with a wrist actigraphy or ActTrust. ActTrust generates amplitude (peak or maximum of the curve, with a lower amplitude indicating a less rhythmic rhythm).
Circadian Activity Rhythms - Acrophase | Up to 14 months
  Circadian Activity Rhythms (CAR) will be recorded with a wrist actigraphy or ActTrust. ActTrust generates acrophase (time of day of the peak activity, with a later time indicating more phase-delay).
Circadian Activity Rhythms - Mesor | Up to 14 months
  Circadian Activity Rhythms (CAR) will be recorded with a wrist actigraphy or ActTrust. ActTrust generates mesor (half-way between minimum and maximum of the curve, a circadian rhythm-adjusted mean of the daily activity).

CONTACTS AND LOCATIONS:
Overall Officials: Heiddis Valdimarsdottir, PhD, Principal Investigator — Reykjavik University; Birna Baldursdottir, PhD, Study Chair — Reykjavik University; Hannah R Sigurdardottir Tobin, MSc, Study Director — University of Reykjavík
Locations (1):
- Reykjavik University, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ancoli-Israel S, Liu L, Marler MR, Parker BA, Jones V, Sadler GR, Dimsdale J, Cohen-Zion M, Fiorentino L. Fatigue, sleep, and circadian rhythms prior to chemotherapy for breast cancer. Support Care Cancer. 2006 Mar;14(3):201-9. doi: 10.1007/s00520-005-0861-0. Epub 2005 Jul 12. PMID 16010529
- [Background] Bower JE. Behavioral symptoms in patients with breast cancer and survivors. J Clin Oncol. 2008 Feb 10;26(5):768-77. doi: 10.1200/JCO.2007.14.3248. PMID 18258985
- [Background] Merriman JD, Von Ah D, Miaskowski C, Aouizerat BE. Proposed mechanisms for cancer- and treatment-related cognitive changes. Semin Oncol Nurs. 2013 Nov;29(4):260-9. doi: 10.1016/j.soncn.2013.08.006. PMID 24183157
- [Background] Wu LM, Amidi A, Valdimarsdottir H, Ancoli-Israel S, Liu L, Winkel G, Byrne EE, Sefair AV, Vega A, Bovbjerg K, Redd WH. The Effect of Systematic Light Exposure on Sleep in a Mixed Group of Fatigued Cancer Survivors. J Clin Sleep Med. 2018 Jan 15;14(1):31-39. doi: 10.5664/jcsm.6874. PMID 29198295
- [Derived] Aspelund SG, Halldorsdottir T, Agustsson G, Tobin HRS, Wu LM, Amidi A, Johannsdottir KR, Lutgendorf SK, Telles R, Daly HF, Sigurdardottir K, Figueiro MG, Redd WH, Valdimarsdottir HB, Baldursdottir B. The Effects of Light Therapy on Cognitive Function and Stress in Women With Breast Cancer Before Systemic Treatment. Cancer Med. 2025 Nov;14(22):e71412. doi: 10.1002/cam4.71412. PMID 41275449
- [Derived] Aspelund SG, Halldorsdottir T, Agustsson G, Sigurdardottir Tobin HR, Wu LM, Amidi A, Johannsdottir KR, Lutgendorf SK, Telles R, Daly HF, Sigurdardottir K, Valdimarsdottir HB, Baldursdottir B. Biological and psychological predictors of cognitive function in breast cancer patients before surgery. Support Care Cancer. 2024 Jan 8;32(1):88. doi: 10.1007/s00520-023-08282-5. PMID 38185720